CLINICAL TRIAL: NCT02417649
Title: Sublingual Administration of a Polyvalent Mechanical Bacterial Lysate in Patients With Moderate, Severe or Very Severe COPD According to GOLD Classification: a Multicenter, Double Blind, Randomized, Controlled, Phase IV Study
Brief Title: Advanced Immunological Approach in COPD Exacerbation
Acronym: AIACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lallemand Pharma AG (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PIRRI/CT/001
Record Dates: First submitted 2013-10-14; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ismigen (Experimental): Treatment over 3 successive months. One sublingual tablet every day on the first ten days of each month, followed by twenty days of rest.
  Interventions: Biological: Ismigen
- Placebo (Placebo Comparator): Treatment over 3 successive months. One sublingual tablet every day on the first ten days of each month, followed by twenty days of rest.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — 1. The placebo will be administered for a period of three months. The first ten days of each month, one tablet per day will be given. The tablet will be melted under the tongue. After the ten day therapy, a twenty day of rest will be provided. Then the second and the third month the administration schedule will be identical.
  2. Three months of rest, according to the indications, will be allowed.
  3. A second cycle (the same as point 1.) will be performed
  4. A second three month rest (according to point 2.) will be provided.
  Arms: Placebo
Biological: Ismigen — 1. The tablet will be administered for a period of three months. The first ten days of each month, one tablet per day will be given. The tablet will be melted under the tongue. After the ten day therapy, a twenty day of rest will be provided. Then the second and the third month the administration schedule will be identical.
  2. Three months of rest, according to the indications, will be allowed.
  3. A second cycle (the same as point 1.) will be performed
  4. A second three month rest (according to point 2.) will be provided.
  Arms: Ismigen

SUMMARY:
Chronic obstructive pulmonary disease (COPD) are characterized by frequent relapses, often resulting from common bacterial infections. Enhancing the immune response in these patients may decrease the frequency of these relapses. The use of a mechanic Polyvalent Bacterial Lysate (PMBL, Ismigen, 13 bacterial strains)may enhance the immune response and therefore help significantly to the control of relapse in these patients.

In the current study the effect of the administration of the PBML to patients older than 40 years, with moderate, severe or very severe COPD, in good or discrete physical condition on the number of relapses in an observation period of 12 months. In addition, the effect of the PMBL on the duration of the interval between relapses, on relapse symptoms, on the use of other drugs, on the number of days of absence of work, on the number of hospitalizations and duration thereof and on potential toxicity of the treatment.

DETAILED DESCRIPTION:
Ancillary Study at the center of Genoa:

To investigate in a subgroup of patient, taking part in the AIACE study, the ability of PMBL to induce an Ig response, to modify the NK blood pattern, and to modulate inflammatory parameters (e.g. CRP).

Material & Methods:

30 patients who were enrolled at the Respiratory Department of Genoa University during the AIACE trial and double blind randomly treated with bacterial lysate or placebo, will participate in this ancillary study.

A further informed consent to participate in this laboratory trial will be requested to the patient besides the already ethical procedure approved for the AIACE study.

In order to assess the enhancement of the concentration of salivary antibodies, a sample of salivary fluid (SF) will be collected at day 0 using Salivette (Starsted, Germany, used according to the manufacture's instructions) and stored frozen until assayed. Then, treatment with PMBL will be carried out for ten days. After twenty-day rest (day 30), at the end of first treatment course (day 90) at the beginning and at the end of the second drug course (day 180, 210) and at the end of the study (day 360), a SF sample will be collected and stored frozen.

Besides the AIACE laboratory procedure already approved, a further blood sample (6 glass tubes) will be collected for peripheral NK blood phenotyping and CRP dosage.

Purified NK cells will obtained from peripheral blood sample at time 0, 90 and 360 by negative selection by using the NK cell isolation Kit (Miltenyi Biotech, Bergisch Gladbach - Germany) following the manufacturer instructions. The NK cell populations are assessed for purity and only those homogeneously displaying CD3-CD14-CD15-CD19- phenotype are selected.

Cells obtained as above described will be analyzed (time t0) by flow cytometry using the following mAbs: anti-CD3, anti-CD56, anti-NKp30, anti-NKp46, anti-NKp44, anti-NKG2D, anti-CD158B1/B2j, anti-KIR p70, anti-CD159A , anti-CD226 (Immunotech -Marseille, France).

In order to assess the efficacy of PMBL on systemic inflammation CRP will be evaluated at day 0 90 and 360. Finally, special T cell subpopulations, such as regulatory T cells, will be assayed on collected samples, together with the concentration of circulating chemokines, cytokines and inflammation-related molecules using a specific immunobeads and flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented moderate, severe and very severe COPD
* Age greater than or equal to 40 years.
* Female patient must be non-lactating and of non-childbearing potential, surgically sterile, or using effective contraception.
* Patients must have WHO performance status of 0, 1 or 2.
* Patients must have adequate hematological, renal and liver function as defined by laboratory values below performed within 14 days, inclusive, prior to study randomization.
* Smokers, ex-smokers can be included but the smoking status is acquired and accurately recorded
* Absolute neutrophil count (ANC) ≥ 2.0 x 109/l.
* Platelet count ≥ 100 x 109/l.
* Hemoglobin ≥ 10 g/dl (> 6.2 mmol/l).
* Urea and serum creatinine <1.5 times upper limit of laboratory normal (ULN).
* Total serum bilirubin <1.5 times ULN.
* ALAT or ASAT <5 times ULN.
* Alkaline phosphatase <5 times ULN.
* Gammaglutamyltransferase (GGT) <5 times ULN.
* LDH <5 times ULN.
* Before patient randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Patients who had received any prior antineoplastic drug therapy or immunosuppressive drugs.
* Patients under continuous treatment with systemic steroids.
* Presence of severe cardiac disease including uncontrolled angina pectoris and myocardial infarction within 6 months, uncontrolled high blood pressure.
* Presence of severe respiratory disease as identified from spirometry and/or chest X ray.
* Presence of any other uncontrolled severe medical condition including active gastroduodenal ulcer, alcohol disorders ( hepatitis, Korsakoff syndrome..), diabetes, active or uncontrolled infection, evolutive intracranial hypertension"
* Patients pregnant or nursing at the beginning of the study.
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To demonstrate the clinical efficacy of Ismigen in patients with moderate, severe and very severe COPD (M/S/VS-COPD) according to GOLD classification, in terms of reduction of the number of exacerbations in a 12 month observation period. | 1 year

SECONDARY OUTCOMES:
Effect of Ismigen on the interval between each exacerbation. | 1 year
Effect of Ismigen on disease symptoms (fever, dyspnoea). | 1 year
Ability of Ismigen to reduce the use of other drugs (antibiotics, antinflammatory drugs, bronchodilators, mucolytics, etc.) in patients with documented M/S/VS-COPD. | 1 year
Ability of Ismigen to reduce the number of days of absence from work in patients with documented M/S/VS-COPD. | 1 year
Number of patients with adverse events as a measure of safety and tolerabiity. | 1 year
Impact on quality of life assessed with a generic health survey (SF-12) and a specific (CCIQ) instrument. | 1 year
Ability of Ismigen (PMBL) to induce immunological and inflammatory modulatory responses | 1 year
  Ancillary study in a subgroup of patient from the AIACE study, the measure the ability of PMBL to induce an Ig response, to modify the NK blood pattern, and to modulate inflammatory parameters (e.g. CRP).
  30 patients who were enrolled at the Respiratory Department of Genoa University during the AIACE trial and double blind randomly treated with bacterial lysate or placebo, will participate in this ancillary study.
Effect of Ismigen on the number of hospitalizations. | 1 year
Effect of Ismigen on the duration of hospitalizations. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Walter Canonica, Prof. MD, Principal Investigator — University of Genova, Genova, Italy
Locations (13):
- Italy (13):
  - Pneumology Department - San Paolo Hospital, Milan, Milan
  - Respiratory Physiopatology and Pneumology Unit, Di Circolo Predabissi-Melegnano hospital, Vizzolo Predabissi, MI
  - Respiratory and Pulmonary desease Unit - IRCCS San Matteo, Pavia, Pavia
  - Specialistic Rehabilitation (Pneumolgi Unit),"Carlo Mira" hospital, Casorate Primo, PV
  - Rehabilitation Pneumology Unit, IRCCS San Raffaele Pisana, Rome, RM
  - Respiratory Clinical Pharmacology, Department of Internal Medicine, Tor Vergata Hospital, Rome, RM
  - Broncopneumology and Allergology Unit, Abbiategrasso hospital, Abbiategrasso
  - Respiratory Physiopatology Unit, Mellino Mellini hospital, Chiari
  - Pneumology Unit, Cremona hospital, Cremona
  - Allergy and Respiratory Diseases Clinic, San Martino hospital, Genova
  - Pneumology Unit, San Gerardo hospital, Monza
  - Complex structure of Pulmonary Allergy, Cardarelli hospital, Naples
  - Complex structure of Pulmonary Rehabilitation, Cardarelli hospital, Naples